CLINICAL TRIAL: NCT02303041
Title: An Open-Label Pilot Study to Evaluate the Efficacy and Safety of a Combination Treatment of Sonidegib (LDE225) and Buparlisib (BKM120) For the Treatment of Advanced Basal Cell Carcinomas
Brief Title: Pilot Study of Sonidegib and Buparlisib in Treating Patients With Advanced or Metastatic Basal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Anne Chang (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Anne Chang, Associate Professor of Dermatology, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-29839; NCI-2014-02200 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SKIN0020 (Other: OnCore); NCT02303041 (Registry Identifier: Stanford University)
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Results first posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Carcinoma, Basal Cell; Recurrent Skin Cancer; Skin Neoplasms; Basal Cell Nevus Syndrome
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms; Basal Cell Nevus Syndrome | interventions — NVP-BKM120; sonidegib

STUDY DESIGN:
Intervention Model Description: Cohort assignment based on disease status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BCC Smoothened inhibitor-naive (Experimental): Participants with locally advanced or metastatic basal cell carcinoma (BCC) and naive to treatment with Smoothened inhibitors receive sonidegib and buparlisib in repeating 28-day cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Buparlisib; Drug: Sonidegib
- BCC refractory or relapsed after Smoothened inhibitor (Experimental): Participants with locally advanced or metastatic basal cell carcinoma (BCC) that is refractory or relapsed after treatment with Smoothened inhibitors receive sonidegib and buparlisib in repeating 28-day cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Buparlisib; Drug: Sonidegib

INTERVENTIONS:
Drug: Buparlisib — Administered orally at starting dose of 80 mg/day
  Other Names: BKM120; PI3K inhibitor BKM120
Drug: Sonidegib — Administered orally at starting dose of 200 mg/day
  Other Names: Sonidegib phosphate; Odomzo; Erismodegib; LDE225

SUMMARY:
This pilot trial studies how well sonidegib and buparlisib work in treating patients with basal cell carcinoma that has spread to other places in the body. Sonidegib and buparlisib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Estimate the overall response rate (ORR) of sonidegib (erismodegib) in combination with buparlisib (hereby referred to as "LB therapy") for patients with locally advanced or metastatic basal cell carcinoma (BCC) in Smoothened inhibitor-naive patients (Cohort 1) and those whose disease is refractory or relapsed on Smoothened inhibitor monotherapy (Cohort 2).

NOTE: This study does not compare the treatment effect between these 2 dissimilar participant groups.

SECONDARY OBJECTIVES:

* Estimate the median duration of response, on or after LB therapy.
* Assess the safety and tolerability of LB therapy.
* Assess the histopathologic effect of LB therapy in tumor biopsies obtained at baseline and following 12 weeks of treatment.
* Assess the effect of LB therapy on gene expression including Hedgehog pathway and phosphatidylinositol 3-kinase (PI3K) pathways.
* Assess correlation between gene mutations in Smoothened, suppressor of fused homolog (Sufu), patched (PTCH), glioma-associated oncogene homolog (Gli)1, 2 and gene expression profiles and response to LB therapy.

OUTLINE:

Patients receive sonidegib orally (PO) once daily (QD) and buparlisib PO QD on days 1 to 28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months.

ELIGIBILITY:
INCLUSION CRITERIA:

* Able to understand and sign informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Metastatic BCC, histologic confirmation of distant BCC metastasis
* Metastatic disease, target lesion must be measurable using computed tomography (CT) or magnetic resonance imaging (MRI)
* Locally advanced BCC are required to have disease that is considered inoperable due to significant functional compromise or to have a medical contraindication to surgery
* Nevoid BCC syndrome (Gorlin syndrome) may enroll in this study but must meet the criteria for locally advanced or metastatic disease listed above
* COHORT 2 ONLY: A Smoothened inhibitor must have been previously administered as monotherapy
* Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
* Platelets ≥ 80 x10^9/L
* Hemoglobin (Hb) > 9 g/dL or values ≥ lower limit of normal (LLN) for site-specific lab
* Total calcium (corrected for serum albumin) within normal limits (biphosphonate use for malignant hypercalcemia control is not allowed)
* Magnesium ≥ the lower limit of normal
* Potassium within normal limits for the institution
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within normal range [or ≤ 3.0 x upper limit of normal (ULN) if liver metastases are present]
* Serum bilirubin within normal range (or ≤ 1.5 x ULN if liver metastases are present; or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in patients with well-documented Gilbert Syndrome)
* Serum creatinine ≤ 1.5 x ULN or 24-hour clearance ≥ 50 mL/min
* Serum amylase ≤ ULN
* Serum lipase ≤ ULN
* Fasting plasma glucose ≤ 120 mg/dL (6.7 mmol/L)
* Negative serum pregnancy test within 72 hours before starting study treatment in women with childbearing potential
* International normalized ratio (INR) ≤ 2

EXCLUSION CRITERIA:

* Prior treatment with a P13K inhibitor
* Known hypersensitivity to buparlisib or to its excipients
* Untreated brain metastases are excluded; however, patients with metastatic central nervous system (CNS) tumors may participate in this trial, if the patient is > 4 weeks from therapy completion (including radiation and/or surgery), is clinically stable at the time of study entry and is not receiving corticosteroid therapy
* Acute or chronic liver, renal disease or pancreatitis
* Baseline creatinine kinase (CK) > ULN
* The following mood disorders as judged by the Investigator or a psychiatrist, or as a result of patient's mood assessment questionnaire:

  * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others)
  * ≥ Common Terminology Criteria for Adverse Events (CTCAE) grade 3 anxiety
  * Meets the cut-off score of ≥ 12 in the Patient Health Questionnaire (PHQ)-9 or a cut-off of ≥ 15 in the Generalized Anxiety Disorder 7-item (GAD-7) mood scale, respectively, or selects a positive response of "1, 2, or 3" to question number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9)
* Diarrhea ≥ CTCAE grade 2
* Active cardiac disease including any of the following:

  * Left ventricular ejection fraction (LVEF) < 50% as determined by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO)
  * QTc > 450 msec on screening electrocardiogram (ECG) (using the QTcF formula)
  * Angina pectoris that requires the use of anti-anginal medication
  * Ventricular arrhythmias except for benign premature ventricular contractions
  * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
  * Conduction abnormality requiring a pacemaker
  * Valvular disease with document compromise in cardiac function
  * Symptomatic pericarditis
* Patient has a history of cardiac dysfunction including any of the following:

  * Myocardial infraction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function
  * History of documented congestive heart failure (New York Heart Association functional classification 3-4)
  * Documented cardiomyopathy
* Patient has poorly controlled diabetes mellitus [defined as hemoglobin A1C (HgA1c) > ULN], steroid-induced diabetes mellitus, or insulin dependent diabetes mellitus
* Other concurrent severe and/or uncontrolled concomitant medical conditions (eg, active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol
* Significant symptomatic deterioration of lung function; if clinically indicated, pulmonary function tests including measures of predicted lung volumes, diffusing capacity of the lung for carbon monoxide (DLco), oxygen (O2) saturation at rest on room air should be considered to exclude pneumonitis or pulmonary infiltrates
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of buparlisib (eg, ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection); patients with unresolved diarrhea will be excluded as previously indicated
* Patients who have been treated with any hematopoietic colony-stimulating growth factors (eg, filgrastim (granulocyte-colony stimulating factor, G-CSF), sargramostim (granulocyte-macrophage colony-stimulating factor, GM-CSF) ≤ 2 weeks prior to starting study drug; erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued
* Patients who are currently receiving treatment with medication with a known risk to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug
* Patients receiving chronic treatment with steroids or another immunosuppressive agent

  * Note: topical applications (eg, rash), inhaled sprays (eg, obstructive airways diseases), eye drops or local injections (eg, intr-articular) are allowed; patients with previously treated brain metastases, who are on stable low dose corticosteroids treatment (eg, dexamethasone 2 mg/day, prednisolone 10 mg/day) for at least 14 days before start of study treatment are eligible
* Patients who have taken herbal medications and certain fruits within 7 days prior to starting study drug; herbal medications include, but are not limited to St. John's Wort, Kava, ephedra (ma huang), dehydroepiandrosterone (DHEA), gingko biloba, yohimbe, saw palmetto, and ginseng; fruits include the cytochrome P450, family 3, subfamily A (CYP3A) inhibitors Seville oranges, grapefruit, pummelos, or exotic citrus fruits
* Patients who are currently treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug; please note that co-treatment with weak inhibitors of CYP3A is allowed
* Patients who have received chemotherapy or targeted anticancer therapy ≤ 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug must recover to a grade 1 before starting the trial
* Patients who have received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) ≤ 5 effective half lives prior to starting study drug or who have not recovered from side effects of such therapy
* Use of statin drugs or other medications known to associate with rhabdomyolysis; these drugs must be discontinued at enrollment
* Patients who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who are currently taking therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulant; low molecular weight heparin is allowed
* Women who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control; double barrier contraceptives must be used through the trial by both sexes; oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study; women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (ie, who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test ≤ 72 hours prior to initiating treatment

  * Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (eg, age appropriate, history of vasomotor symptoms) or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone (FSH) levels > 40 mIU/mL (for US only: and estradiol < 20 pg/mL) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least 6 weeks prior; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
  * Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during the study and through 20 months after the final dose of study treatment; for males with partners with childbearing potential, highly effective contraception is required for 6 months; the highly effective contraception is defined as either:

    * True abstinence: when this is in line with the preferred and usual lifestyle of the subject; periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate); for female subjects on the study, the vasectomized male partner should be the sole partner for that patient
    * Use of a combination of any two of the following (a+b):

      * a. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
      * b. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
  * Oral contraception, injected or implanted hormonal methods are not allowed
  * Fertile males, must use highly effective (double barrier) methods of contraception (eg, spermicidal gel plus condom) for the entire duration of the study, and continuing using contraception and refrain from fathering a child for 6 months following the study drug; a condom is required to be used also by vasectomized men as well as during intercourse with a male partner in order to prevent delivery of the study treatment via seminal fluid; female partner of male study subject should use highly effective contraception during dosing of any study agent and for 16 weeks after final dose of study therapy
  * Note: hormonal contraception methods (eg, oral, injected, implanted) are not allowed
  * Note: woman are considered post-menopausal and not child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (eg, age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 20 pg/mL or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago; in the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential
* Known diagnosis of human immunodeficiency virus (HIV) infection, hepatitis B or hepatitis C
* History of another malignancy within 3 years, except cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix
* Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Lynn Chang, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tran DC, Moffat A, Brotherton R, Pague A, Zhu GA, Chang ALS. An exploratory open-label, investigator-initiated study to evaluate the efficacy and safety of combination sonidegib and buparlisib for advanced basal cell carcinomas. J Am Acad Dermatol. 2018 May;78(5):1011-1013.e3. doi: 10.1016/j.jaad.2017.11.031. Epub 2017 Nov 23. No abstract available. PMID 29175429

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BCC Smoothened Inhibitor-naive | BCC Refractory or Relapsed After Smoothened Inhibitor
Started | 4 | 6
Completed | 3 | 4
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BCC Smoothened Inhibitor-naive | BCC Refractory or Relapsed After Smoothened Inhibitor | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 6
  >=65 years | 2 | 2 | 4
Age, Continuous [Median (Standard Deviation); unit: years] | 72.3 (20.9) | 60.7 (8.01) | 61.2 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 6 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Response was assessed by the Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria, and reported as overall response rate (ORR), comprised of the sum of complete response (CR) rate and partial response (PR) rate.
  * Complete Response (CR) = Disappearance of all target lesions
  * Partial Response (PR) = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Overall Response (OR) = CR + PR
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | BCC Smoothened Inhibitor-naive | BCC Refractory or Relapsed After Smoothened Inhibitor
Number analyzed (Participants) | 3 | 4
Participants | 0 | 1

2. Secondary Outcome: Median Duration of Response
Description: Response per the Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 criteria was monitored for duration of response (DOR)
  * Complete Response (CR) = Disappearance of all target lesions
  * Partial Response (PR) = ≥ 30% decrease in the sum of the longest diameter of target lesions
  * Overall Response (OR) = CR + PR
  * Progressive disease (PD) = 20% increase in the sum of the longest diameter of target lesions
  * Stable disease (SD) = Small changes that do not meet any of the above criteria
Time Frame: up to 12 weeks
Population: Most participants were not evaluable per protocol.
Measure: Median (Full Range); unit: months
Arm/Group | BCC Smoothened Inhibitor-naive | BCC Refractory or Relapsed After Smoothened Inhibitor
Number analyzed (Participants) | 0 | 1
months |  | 13.8 [13.8 to 13.8]

3. Secondary Outcome: Adverse Event Frequency
Description: Adverse events, graded according to the National Cancer Institute CTCAE version 3.0, are reported by treatment arm in total and by Grade 1 to 5.
Time Frame: Up to 30 days post-treatment
Measure: Number; unit: adverse events
Arm/Group | BCC Smoothened Inhibitor-naive | BCC Refractory or Relapsed After Smoothened Inhibitor
Number analyzed (Participants) | 4 | 6
adverse events
  Grade 1 (mild) | 30 | 43
  Grade 2 (moderate) | 16 | 33
  Grade 3 (severe) | 3 | 5
  Grade 4 (life-threatening) | 0 | 0
  Grade 5 (fatal) | 0 | 0
  All adverse events | 49 | 81

4. Secondary Outcome: Changes in Gene Expression Profiles of BCCs Including Hedgehog Pathway and PI3K Pathways
Description: Immunostaining for the Gli-1; Gli-2; "Patched" (Ptch) ; "Suppressor of Fused" (SuFu); "Smoothened" (Smo)"; and phosphatidylinositol-3-kinase (PI3K) cellular biomarkers were to be contacted at baseline and after 12 weeks of treatment.
Time Frame: Baseline to 2 years
Population: The individual samples were not analyzed for the biomarkers due to the overall small sample size.
Arm/Group | BCC Smoothened Inhibitor-naive | BCC Refractory or Relapsed After Smoothened Inhibitor
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Gene Expression Profiles (Correlation of Particular Gene Expression Profiles and Response to LB Therapy Will be Assessed.)
Description: The gene expression profiles for Gli-1; Gli-2; "Patched" (Ptch) ; "Suppressor of Fused" (SuFu); "Smoothened" (Smo)"; and phosphatidylinositol-3-kinase (PI3K) were to be correlated to the clinical response to therapeutic therapy.
Time Frame: up to 2 years post-treatment
Population: The individual samples were not analyzed for the biomarkers due to the overall small sample size, and thus the correlation of gene expression profile to therapeutic response was not conducted.
Arm/Group | BCC Smoothened Inhibitor-naive | BCC Refractory or Relapsed After Smoothened Inhibitor
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | BCC Smoothened Inhibitor-naive | BCC Refractory or Relapsed After Smoothened Inhibitor
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/6
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCC Smoothened Inhibitor-naive (N=4) | BCC Refractory or Relapsed After Smoothened Inhibitor (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Alanine aminotransferase increase (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCC Smoothened Inhibitor-naive (N=4) | BCC Refractory or Relapsed After Smoothened Inhibitor (N=6)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis, oral (Gastrointestinal disorders) | 1 (1) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders-Other, Abdominal cramps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increase (Investigations) | 1 (1) | 1 (2)
Alanine aminotransferase increase (Investigations) | 1 (1) | 1 (1)
Creatine phosphokinase increase (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0)
Muscle spasm or cramps (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 2 (2) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (4)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 4 (4) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin & subcutaneous tissue disorders-others, Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1)
Flu-like symptoms (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 6 (7)
Eye disorders-Others, change in vision (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 2 (2) | 0 (0)
Ear pain (Otalgia) (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neoplasms - Other, Malignant, skin, squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasms - Other, Malignant, skin, basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps)-Others, Unspecified, skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Other, bleeding (shoulder) (Blood and lymphatic system disorders) | 1 (3) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 3 (4)
Surgical and medical procedures-others, Moh's surgery for SCC (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures (Surgical and medical procedures) | 0 (0) | 1 (1)
Surgical and medical procedures-others Cyst Removal (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT02303041/Prot_SAP_000.pdf